CLINICAL TRIAL: NCT03882021
Title: High-Density (HD) Wave Mapping in Subjects With Atrial Fibrillation as a Predictor of Recurrence After a Single Ablation Procedure Using a PVI-Only Strategy
Acronym: WAVE-MAP AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABT-CIP-10275
Record Dates: First submitted 2019-03-07; First posted 2019-03-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Cardiac Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: All subjects enrolled will undergo the same mapping and ablation protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mapping protocol with Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ (GRID) catheter (Other): All patient will undergo a protocol required mapping protocol using the GRID catheter.
  Interventions: Procedure: A specific electrophysiology mapping protocol is applicable with the GRID catheter.

INTERVENTIONS:
Procedure: A specific electrophysiology mapping protocol is applicable with the GRID catheter. — The procedure will be done according to a standard ablation approach. During the electrophysiology study, additional mapping data will be collected to support the study endpoints using the GRID catheter.

SUMMARY:
The aim is to use the Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ to characterize the atrial substrate and develop a model for predicting recurrence rates after a single procedure using a PVI only approach and a contact catheter.

DETAILED DESCRIPTION:
This clinical investigation is intended to characterize the left atrial substrate using the Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ in an HD Wave configuration and correlate different factors with 12-month success after a single ablation procedure using a pulmonary vein isolation (PVI) approach without further substrate modification.

This is a post-market, single-arm, multi-center, prospective interventional study of the Advisor™ HD Grid Mapping Catheter, Sensor Enabled™. This study is aimed at determining correlations between pre-ablation mapping characteristics and outcomes after catheter ablation of atrial fibrillation.

Approximately 300 subjects at up to 20 sites worldwide will be enrolled.

Subjects will be followed until they complete their 12-month visit. Clinical Investigation visits will occur at Baseline (confirmation of eligibility), Index Procedure, 3 months, 6 months, and 12 months. Endpoints will be analyzed when all subjects have completed their 12-month follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Documented atrial fibrillation with planned endocardial ablation procedure
2. Age 18 years or older
3. Able and willing to provide written informed consent prior to any clinical investigation related procedure
4. Able and willing to complete all required study procedures through 12 months

Exclusion Criteria:

1. Long-standing persistent atrial fibrillation defined as continuous AF greater than 12 months in duration
2. Previous ablation or surgery in the left atria
3. Implanted left atrial appendage occluder
4. Implanted mitral or tricuspid valve replacement
5. Implanted cardiac defibrillator (ICD)
6. Participation in another clinical investigation that may confound the results of this study
7. Pregnant or nursing
8. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
9. Life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, Study Director — Abbott
Locations (15):
- Kepler Universitätsklinikum GmbH, Linz, UPR AUS, Austria
- FN U sv. Anny v Brno, Brno, Moravia-Silesia, Czechia
- France (3):
  - CHR de La Reunion - Site du CHFG, Saint-Denis, ILE
  - Hôpital Privé du Confluent, Nantes, Paysdel
  - Médipôle Lyon-Villeurbanne, Villeurbanne, Rhone
- Germany (3):
  - Klinikum Ingolstadt GmbH, Ingolstadt, Bavaria
  - Herz- u. Gefäßzentrum Bad Bevensen, Bad Bevensen, L Saxon
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
- Italy (2):
  - Ospedale San Raffaele, Milan, Lombard
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Universitair Medische Centrum Groningen, Groningen, Netherlands
- Hospital de Santa Cruz, Carnaxide, Lisbon District, Portugal
- Spain (2):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Vall d'Hebron, Barcelona
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A patient was considered enrolled in the clinical investigation from the moment all of the following enrollment criteria were met: the patient provided written informed consent, patient was confirmed to meet all inclusion criteria and none of the exclusion criteria and the mapping catheter was inserted into the subject's vasculature. If the procedure was cancelled or aborted after consent but prior to the mapping catheter insertion, the subject was withdrawn prior to enrollment.
Groups:
- Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter: All patients will undergo a protocol required mapping protocol using the Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ (GRID) catheter.
  A specific electrophysiology mapping protocol is applicable with the GRID catheter. The procedure will be done according to a standard ablation approach. During the electrophysiology study, additional mapping data will be collected to support the study endpoints using the GRID catheter.
Period: Consent
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Started | 303
Completed | 303
Not Completed | 0
Period: Enrollment
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Started | 303
Completed | 300
Not Completed | 3
Not completed — Procedure aborted/cancelled | 2
Not completed — HD Grid catheter not introduced into patient | 1
Period: Enrollment to 3-Month
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Started | 300
Completed | 291
Not Completed | 9
Not completed — Death | 1
Not completed — Operator not able to achieve PVI | 4
Not completed — Missed Visit | 4
Period: 3-Month to 6-Month Visit
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Started | 295
Completed | 294
Not Completed | 1
Not completed — Missed Visit | 1
Period: 6-Month to 12-Month Visit
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Started | 295
Completed | 287
Not Completed | 8
Not completed — Death | 1
Not completed — Missed Visit | 7

BASELINE CHARACTERISTICS:
Groups:
- Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter: All patients will undergo a protocol required mapping protocol using the Advisor™ HD Grid Mapping Catheter, Sensor Enabled™(GRID) catheter.
  A specific electrophysiology mapping protocol is applicable with the GRID catheter. The procedure will be done according to a standard ablation approach. During the electrophysiology study, additional mapping data will be collected to support the study endpoints using the GRID catheter.
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 211
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 9
  Netherlands | 13
  Czechia | 68
  Italy | 43
  United Kingdom | 10
  France | 74
  Portugal | 5
  Germany | 59
  Spain | 12
  Israel | 2
  Poland | 5
Height [Mean (Standard Deviation); unit: inches] | 68.5 (3.8)
Weight [Mean (Standard Deviation); unit: lbs] | 189.3 (37.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (4.6)
New York Heart Association (NYHA) [Count of Participants; unit: Participants] — NYHA classifies patients' heart failure into one of four categories based on limitations of physical activity. Class I is no limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitations, or shortness of breath. Class IV is symptoms of heart failure at rest. Any physical activity causes further discomfort. Population: Only evaluated for subjects with a history of heart failure.
  Participants
    number analyzed (Participants) | 82
    I | 13
    II | 48
    III | 16
    IV | 0
    Not evaluated | 5
History of heart failure [Count of Participants; unit: Participants] | 82
Transthoracic Echocardiogram (TTE) performed [Count of Participants; unit: Participants] | 296
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] — Population: Only evaluated in subjects with available data.
  %
    number analyzed (Participants) | 288
    (all) | 57.4 (8.5)
Evidence of left ventricular hypertrophy [Count of Participants; unit: Participants] — Population: Only evaluated in subjects in which a TTE was performed.
  Participants
    number analyzed (Participants) | 296
    (all) | 47
Evidence of hypertrophic cardiomyopathy [Count of Participants; unit: Participants] — Population: Only evaluated in subjects in which a TTE was performed.
  Participants
    number analyzed (Participants) | 296
    (all) | 6
History of Hypertension [Count of Participants; unit: Participants] | 179
Diabetes [Count of Participants; unit: Participants] | 34
Coronary Artery Disease [Count of Participants; unit: Participants] | 33
Subject has a pacemaker [Count of Participants; unit: Participants] | 5
Valvular Heart Disease [Count of Participants; unit: Participants] | 69
Stroke/Transient Ischemic Attack (TIA)/Thromboembolism [Count of Participants; unit: Participants] | 23
Paroxysmal Atrial Fibrillation (less than 7 days) [Count of Participants; unit: Participants] | 113
Early Persistent Atrial Fibrillation (7 days - 3 months) [Count of Participants; unit: Participants] | 86
Non-Early Persistent Atrial Fibrillation (3-12 months) [Count of Participants; unit: Participants] | 101
Typical Atrial Flutter [Count of Participants; unit: Participants] | 47
Class I/III Anti-arrhythmic drug (AAD) (currently taking/previously taken) [Count of Participants; unit: Participants] | 186

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With One-year Success
Description: Defined as freedom from atrial fibrillation, atrial flutter and atrial tachycardia after removal from the antiarrhythmic drug therapy as assesses from the end of the 3-month blanking period to 12 months following a single ablation procedure. Kaplan-Meier survival analysis will be conducted to analyze time-to-event variables.
Time Frame: the end of the 3-month blanking period to 12 months following a single ablation procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
percentage of participants | 57.2 [51.2 to 62.8]
Statistical Analysis 1: Comparison: Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter; Test type: Other; Kaplan Meier Survival Estimate = 57.2, 95% CI 2-sided [51.2 to 62.8], Standard Error of Mean 3.0 — Kaplan-Meier estimate of freedom from recurrence after removal from AAD at one year

2. Other Pre Specified Outcome: Percentage of Subjects With Freedom From Symptomatic AF/AFL/AT After Removal From Antiarrhythmic Drug Therapy
Description: Percentage of participants with freedom from symptomatic atrial fibrillation/atrial flutter/atrial tachycardia rafter removal from AADs. Kaplan-Meier survival analysis was conducted to analyze time-to-event variables.
Time Frame: the end of the 3-month blanking period to 12 months after initial ablation procedure
Measure: Number; unit: percentage of participants
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
percentage of participants | 61.7
Statistical Analysis 1: Comparison: Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter; Test type: Other — Kaplan Meier Estimate of freedom from symptomatic recurrence; Kaplan-Meier Survival Estimate = 61.7, 95% CI 2-sided [55.8 to 67.1], Standard Error of Mean 2.9 — Kaplan-Meier estimate of freedom from symptomatic AF/AFL/AT recurrence after removal from AAD

3. Other Pre Specified Outcome: Percentage of Subjects With Single Procedure Clinical Success
Description: Single procedure clinical success was defined as freedom from symptomatic atrial fibrillation, atrial flutter and atrial tachycardia without a new or increased dose of class I or III antiarrhythmic drug. Kaplan-Meier survival analysis was conducted to analyze time-to-event variables.
Time Frame: the end of the 3-month blanking period to 12 months following the initial ablation procedure
Measure: Number; unit: percentage of participants
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
percentage of participants | 79.4
Statistical Analysis 1: Comparison: Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter; Test type: Other — Kaplan Meier estimate of single procedure clinical success; Kaplan-Meier Survival Estimate = 79.4, 95% CI 2-sided [74.2 to 83.6], Standard Error of Mean 2.4 — Kaplan-Meier estimate of freedom from symptomatic AF/AFL/AT without new or increased dose of Class I/III AAD at one year

4. Other Pre Specified Outcome: Percentage of Subjects With Freedom From AF/AFL/AT
Description: Freedom from atrial fibrillation, atrial flutter and atrial tachycardia recurrence. Kaplan-Meier survival analysis was conducted to analyze time-to-event variables.
Time Frame: the end of the 3-month blanking period to 12 months following the initial ablation procedure
Measure: Number; unit: percentage of participants
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
percentage of participants | 75.5
Statistical Analysis 1: Comparison: Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter; Test type: Other — Kaplan Meier estimate of freedom from AF/AFL/AT; Kaplan Meier Survival Estimate = 75.5, 95% CI 2-sided [69.9 to 80.1], Standard Error of Mean 2.6 — Kaplan Meier estimate of freedom from AF/AFL/AT at 12 months

5. Other Pre Specified Outcome: Number of Subjects With Acute Procedural Success
Description: Defined as electrical isolation of all pulmonary veins. The data will be summarized with subject counts and percentages/rates.
Time Frame: During procedure, an average of 160 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
Participants | 296

6. Other Pre Specified Outcome: Number of Subjects With Arrhythmia Recurrence
Description: Rates of recurrence not due to PVI gap for subjects with repeat electrophysiology studies. The data will be summarized with subject counts and percentages/rates.
Time Frame: 12 months
Population: Subjects with repeat electrophysiology studies in which treatment other than ablation of isthmus dependent atrial flutter was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 25
Participants | 3

7. Other Pre Specified Outcome: Left Atrium (LA) Information: LA Volume (LAV)
Description: LA volume will be summarized with the mean with standard deviation.
Time Frame: Baseline
Population: Number of subjects in which LAV was measured.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 151
mL | 68.5 (31.9)

8. Other Pre Specified Outcome: Left Atrium (LA) Information: LA Diameter (LAD)
Description: LA diameter will be summarized with the mean with standard deviation.
Time Frame: Baseline
Population: Includes subjects in which LAD was measured
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 226
mm | 43.1 (12.2)

9. Other Pre Specified Outcome: Reportable Adverse Events
Description: Number of adverse events, including any device-, procedure-, or death-related events (serious or non-serious).
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
Number analyzed (Participants) | 300
events | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter
All-Cause Mortality (participants affected / at risk) | 2/300
Serious Adverse Events (participants affected / at risk) | 8/300
Other Adverse Events (participants affected / at risk) | 7/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter (N=300)
Arrhythmia New (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Valve insufficiency (Cardiac disorders) | 1 (1)
Neurological symptoms (General disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mapping Protocol With Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ Catheter (N=300)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Bleeding/Anemia (Blood and lymphatic system disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pulmonary Vein Stenosis (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Dyspnea at exercise (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results will be made as a joint multi-center publication with investigators from all sites contributing data. Institutions may publish data and results individually from its site after any of the following (1) a multi-center publication is published, (2) no multicenter publication is submitted within eighteen months after closures of the Study at all sites or (3) sponsor confirms in writing there will be no multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT03882021/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT03882021/SAP_001.pdf